CLINICAL TRIAL: NCT06150365
Title: Single Arm Clinical Study on the Safety and Efficacy of Personalized KSX01-TCRT in Patients With Advanced Solid Tumors
Brief Title: Personalized KSX01-TCRT in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSX01-R08-102
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Refractory Solid Tumors; Relapsed Solid Tumors

STUDY DESIGN:
Intervention Model Description: KSX01-TCRT cell therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR-T cells (Experimental): KSX01-TCRT cell therapy
  Interventions: Biological: KSX01-TCRT cell therapy

INTERVENTIONS:
Biological: KSX01-TCRT cell therapy — Patient autologous T cell therapy

SUMMARY:
This trial is a single arm, open phase I clinical study to investigate the safety and efficacy of personalized KSX01-TCRT in patients with advanced solid tumors. This experiment is divided into two parts: the dose increasing stage (Part A) and the dose expanding stage (Part B). For those enrolled in the planned expansion phase, the dose should have passed the safety assessment during the dose escalation phase.

ELIGIBILITY:
Inclusion Criteria:

* Screening period 1- inclusion criteria:

Patients should complete all examinations for screening period 1 within 28 days after signing the informed consent form. Only those who meet the inclusion criteria for this stage can collect fresh tumor tissue, 2-3 archived pathological tissue white slides, and peripheral blood for TCR sequence screening and HLA typing testing.

1. Volunteer to participate in clinical research; Fully understand this study and voluntarily sign an informed consent form; Willing to follow and capable of completing all testing procedures.
2. Age range from 18 to 70 years old (including boundary values).
3. Solid tumors that have been confirmed by histological or cytological evaluation as incurable or metastatic, and have failed standard treatment or currently have no available standard treatment.
4. Expected survival time>6 months.
5. ECOG score 0 or 1.
6. Having sufficient organ function, defined as follows:

   6.1) Hematology: 6.1.1) Hemoglobin 90 g/L (no blood transfusion received within 14 days prior to examination); 6.1.2) Absolute value of neutrophils 1.5 109/L (did not receive granulocyte colony stimulating factor treatment within 14 days prior to examination); 6.1.3) Platelet count is 100 109/L in the absence of obvious liver lesions (primary or metastatic) (platelet transfusion not received within 14 days before examination), or 75 109/L in the presence of liver lesions (platelet transfusion not received within 14 days before examination); 6.1.4) Absolute lymphocyte count (ALC) 0.7 109/L; 6.2) Liver function: 6.2.1) Total bilirubin (TBIL) ≤ 1.5 in the absence of obvious liver lesions (primary or metastatic) × Upper limit of normal (ULN), subjects with liver lesions or Gilbert disease ≤ 3 × ULN; 6.2.2) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (liver metastasis or liver cancer subjects can be ≤ 5 × ULN); Alkaline phosphatase (ALP) ≤ 2.5 × ULN (bone metastasis subject, ALP ≤ 5) × ULN); 6.3) Renal function: Creatinine clearance rate ≥ 60 mL/min (Cockcroft Fault formula: [140 age] × Weight [kg] × [0.85, female only]/(72 × Creatinine (mg/dl);

   Subjects with a creatinine clearance rate of<60 mL/min but ≥ 50 mL/min can also be enrolled if all of the following conditions are met:

   Serum creatinine and blood urea nitrogen (BUN) are within the normal range of the research center No clinical evidence showing chronic renal dysfunction (such as acidosis or electrolyte disorders) The urine routine and urine output are within the normal range of the research center Note: It is not recommended to use IL-2 during the treatment period for subjects with a baseline creatinine clearance rate of<60 mL/min.
7. The patient's HLA-I class molecule IHC expression is positive.
8. Patients with tumor lesions that can be collected and can screen out TCR sequences that can be used as drugs can enter the study. If the patient has obtained personalized TCR sequences using previously collected and archived tumor tissue in other studies, they can directly enter screening period 2, but the collection time of the archived tissue should be within one year before signing the informed consent for this study.
9. The patient agrees to receive peripheral monocyte collection after all tests in screening period 1 meet the standards.

   * Screening period 2- inclusion criteria:

After receiving confirmation notification of TCR sequence locking from the partner, or if the patient has obtained their personalized TCR sequence in other studies, they can be arranged to undergo various inclusion evaluations in screening period 2.

The organ function and key examination items of the patient at this stage should not have significant changes compared to the examination results in screening period 1. If the patient's examination results during screening period 2 exceed the following criteria, peripheral monocyte collection should not be performed until the abnormal items return to normal range.

Screening period 2- Routine inclusion criteria

1. Confirmed screening and locking of tumor specific TCR sequences from the patient's own body. For patients who have obtained TCR sequences through other research projects, they should sign an informed consent form for this research project before entering screening period 2.
2. Expected survival time>6 months.
3. ECOG score 0 or 1.
4. Having sufficient organ function, defined as follows:

4.1) Hematology: 4.1.1) Hemoglobin 90 g/L (no blood transfusion received within 14 days prior to examination); 4.1.2) Absolute value of neutrophils is 1.0 109/L (did not receive granulocyte colony stimulating factor treatment within 14 days before the examination); 4.1.3) Platelet count is 75 109/L in the absence of obvious liver lesions (primary or metastatic) (platelet transfusion was not received within 14 days before the examination); 4.1.4) Absolute lymphocyte count (ALC) 0.7 109/L; 4.2) Liver function: 4.2.1) Total bilirubin (TBIL) ≤ 1.5 in the absence of obvious liver lesions (primary or metastatic) × Upper limit of normal (ULN), subjects with liver lesions or Gilbert disease ≤ 3 × ULN; 4.2.2) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (liver metastasis or liver cancer subjects can be ≤ 5 × ULN); Alkaline phosphatase (ALP) ≤ 2.5 × ULN (bone metastasis subject, ALP ≤ 5) × ULN); 4.3) Renal function: Creatinine clearance rate ≥ 60 mL/min (Cockcroft Fault formula: [140 age] × Weight [kg] × [0.85, female only]/(72 × Creatinine (mg/dl);

Subjects with a creatinine clearance rate of<60 mL/min but ≥ 50 mL/min can also be enrolled if all of the following conditions are met:

Serum creatinine and blood urea nitrogen (BUN) are within the normal range of the research center No acidosis or electrolyte disorders The urine routine and urine output are within the normal range of the research center Note: It is not recommended to use IL-2 during the treatment period for subjects with a baseline creatinine clearance rate of<60 mL/min.

4.4) The patient naturally breathes (without assisted oxygen supply) with a basal blood oxygen saturation of>92%.

Agree to accept peripheral monocyte collection. 6) Women of childbearing age who have the ability to conceive have a negative blood pregnancy test within 7 days before the first cell infusion (non fertility: surgical sterilization or at least 2 years after menopause), and the subjects of childbearing age use medically recognized contraceptive measures from the start of research treatment (chemotherapy) to 5 months after the last cell infusion, and no eggs have been retrieved during this period.

7) Male participants are willing to take medically approved contraceptive measures within 5 months after signing the informed consent form and the last cell infusion, and do not donate sperm during this period.

8) According to the iRECIST standard, there is at least one measurable lesion present. The following situations require approval from the researcher:

* During the dose increasing stage, subjects only have evaluable lesions but can evaluate their efficacy through their serum tumor markers;
* The subjects currently do not have measurable lesions, but the researchers have determined that they may develop or become measurable lesions within one month.

  9) The toxicity and adverse reactions caused by frontline treatment should be restored to Grade 1 (excluding clinically insignificant toxicity, such as hair loss caused by chemotherapy).

Exclusion Criteria:

* Screening period 1- Exclusion criteria:

Subjects who meet any of the following criteria shall not participate in this clinical study:

1. The patient has received systemic chemotherapy on line 3 or above:

   Patients can be enrolled during the first line systemic chemotherapy, during the second line systemic chemotherapy period, or after the end of the second line systemic chemotherapy (enrollment time is screening period 2 and meets the standards and receives clearance chemotherapy), but they cannot receive the third line systemic chemotherapy before enrollment:
   * The second and third line systemic chemotherapy is defined as a systematic chemotherapy regimen after the progression of frontline treatment;
   * For patients who complete neoadjuvant chemotherapy in the early stage of their disease, their neoadjuvant chemotherapy regimen can include up to two types of chemotherapy;
   * For patients who meet all other inclusion criteria but have a large number of frontline treatment lines, they can also be included after evaluation and confirmation by the researchers.

   Frontline treatment plans targeting biological agents (such as immune checkpoint inhibitors), small molecule targeted drugs, etc., are not considered as exclusion criteria.
2. Within two years before signing the informed consent, the patient had a medical history of other malignant tumors, except for non melanoma skin cancer, some cancers in situ (such as cervical cancer, bladder cancer, breast cancer), or low-risk prostate cancer.
3. Clinically confirmed liver diseases, including active hepatitis virus infection, alcoholic hepatitis, other types of hepatitis, cirrhosis, and hereditary liver diseases; Among them, the subject's

   * Hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) are positive, and the hepatitis B virus DNA (HBV DNA) in the peripheral blood is higher than the lower detection limit of the research center;
   * HCV-Ab positive and HCV-RNA above the lower detection limit of the research center Patients who can effectively control HBV-DNA and/or HCV-RNA after treatment can also be included in the group after being evaluated and approved by the researcher. HBV-DNA positive subjects should receive hepatitis B treatment after signing the informed consent form and continue to receive KSX01-TCRT infusion for at least 6 months. Such subjects should also monitor their HBV-DNA and hepatitis B related antigen antibodies on Day28 and at each follow-up visit point.
4. History of myocardial infarction, history of cardiac bypass surgery, unstable angina, active atrial fibrillation requiring treatment, symptomatic sinus bradycardia (heart rate<50 beats/min), or other clinically significant heart diseases within 6 months prior to signing the informed consent form.
5. Tumor lesions invading the heart or large blood vessels. The patient has permanent percutaneous nephrostomy, catheterization, bile duct, and other indwelling tubes, except for those that the researchers believe can be removed before gonorrhea clearance.

7) Primary immune deficiency. 8) HIV positive; Active HBV or HCV infection. 9) Received allogeneic stem cell transplantation within 6 months before signing the informed consent form.

10) Prior to signing the informed consent form, CAR T cell therapy or other genetically modified T cell therapy other than this research technique was received.

11) Known allergies to dimethyl sulfoxide (DMSO) or any other cellular formulation components and potential therapeutic drugs used during treatment (such as cyclophosphamide, fludarabine, and tolumab).

12) History of autoimmune diseases, except for the following:

-A history of hypothyroidism and the use of stable thyroid hormone replacement therapy;

-Patient has controllable type 1 diabetes 13) The patient's illness or condition results in their lack of understanding, participation, and/or adherence to this study plan.

14) Any other disease that researchers believe will impair the subject's tolerance to the treatment regimen or significantly increase the risk of complications.

15) Known history of alcohol abuse, psychotropic substance abuse, or drug use. 16) Have a clear history of neurological or mental disorders in the past, such as epilepsy, dementia, schizophrenia, etc.

17) According to the judgment of the researchers, the underlying condition of the subjects may increase their risk of receiving investigational drug treatment, or may cause confusion in the interpretation of toxic reactions and adverse events that may occur.

Other researchers believe that it is not suitable to participate in this study.

* Screening Period 2- Exclusion Criteria

Subjects who meet any of the following criteria shall not undergo peripheral monocyte collection:

1. Before monotherapy, the subject's anti-tumor treatment was not fully eluted (2 weeks or 5 half-lives, whichever is shorter):

   -Except for the following situations: Gonadotropin (GnRH) agonists or antagonists used for the treatment of prostate cancer Hormone replacement therapy or oral contraceptives.
2. Known primary central nervous system (CNS) malignant tumors or symptomatic CNS metastases.

   If the patient is diagnosed with a central nervous system disease and meets the following conditions with the consent of the main researcher, it is not considered an exclusion item:
   * There are measurable or evaluable lesions outside the CNS;
   * No history of intracranial or spinal cord bleeding;
   * There is no need for ongoing or planned corticosteroid treatment within 14 days prior to enrollment;
   * Receiving stable doses of anticonvulsants;
   * No stereotactic radiation or whole brain radiation therapy was received within 14 days prior to enrollment.
3. Women during pregnancy or lactation.
4. Receiving or planning to receive systemic corticosteroid therapy (>5 mg of prednisone or equivalent treatment medication per day) or immunosuppressive drugs within 7 days prior to monotherapy, except for the following:

   * Intranasal, inhalation, topical steroids, or local administration (such as intra articular injection);
   * Physiological doses of systemic steroids as an alternative therapy (such as physiological corticosteroid replacement therapy for adrenal or pituitary dysfunction);
   * Steroids are used as prophylactic drugs for hypersensitivity reactions (such as computed tomography [CT] prophylactic drugs).
5. The first second forced expiratory volume (FEV1)/forced vital capacity (FVC)<70% during lung function examination indicates abnormal lung function.
6. According to the judgment of the researchers, the underlying condition of the subjects may increase their risk of receiving investigational drug treatment, or may cause confusion in the interpretation of toxic reactions and adverse events that may occur.
7. There are severe infections within 2 weeks before single collection. Major surgery (excluding diagnostic surgery) is performed within 4 weeks prior to single collection, or is expected to be performed during the study period. Subjects can be enrolled in planned or ongoing minor surgical procedures, such as establishing venous channels.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Subject safety | about 2 years
  Number of participants with treatment-related adverse events assessed by CTCAE v4.0.
tumor efficacy | about 2 years
  Changes in overall tumor diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Shuhang Wang, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China